CLINICAL TRIAL: NCT00045968
Title: A Phase III Clinical Trial Evaluating DCVax®-L, Autologous Dendritic Cells Pulsed With Tumor Lysate Antigen For The Treatment Of Glioblastoma Multiforme (GBM)
Brief Title: Study of a Drug [DCVax®-L] to Treat Newly Diagnosed GBM Brain Cancer
Acronym: GBM
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Northwest Biotherapeutics (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 020221
Record Dates: First submitted 2002-09-17; First posted 2002-09-19 (Estimated); Last update posted 2022-05-18 (Actual); Status verified 2022-05

CONDITIONS: Glioblastoma Multiforme; Glioblastoma; GBM; Grade IV Astrocytoma; Glioma; Brain Cancer; Brain Tumor
Keywords: oncology; neurology; glioma; brain tumor; brain cancer; glioblastoma multiforme; glioblastoma; newly diagnosed glioblastoma; immunotherapy; dendritic cells; immune therapy; GBM; Brain cancer, primary; tumor vaccine; grade IV astrocytoma; DCVax; Grade IV brain cancer
MeSH Terms: conditions — Glioblastoma; Glioma; Brain Neoplasms; Neoplasms

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- treatment cohort (Active Comparator)
  Interventions: Drug: Dendritic cell immunotherapy
- Placebo Chohort (Placebo Comparator): Autologous PBMC
  Interventions: Drug: Dendritic cell immunotherapy

INTERVENTIONS:
Drug: Dendritic cell immunotherapy — Two intradermal (i.d.) injections of DCVax-L(treatment cohort) or autologous PBMC (placebo cohort) per treatment. Treatments will be given at days 0, 10, 20, and at weeks 8, 16, 32, 48, 72, 96 and 120.
  Other Names: DCVax-L; DCVax; DCVax-Brain

SUMMARY:
The primary purpose of the study is to determine the efficacy of an investigational therapy called DCVax(R)-L in patients with newly diagnosed GBM for whom surgery is indicated. Patients must enter screening at a participating site prior to surgical resection of the tumor. Patients will receive the standard of care, including radiation and Temodar therapy and two out of three will additionally receive DCVax-L, with the remaining one third receiving a placebo. All patients will have the option to receive DCVax-L in a crossover arm upon documented disease progression. (note: DCVax-L when used for patients with brain cancer is sometimes also referred to as DCVax-Brain)

DETAILED DESCRIPTION:
This Phase III trial is designed to evaluate the impact on survival time, as well as safety, in patients following treatment with DCVax(R)-L, an immunotherapy treatment for GBM. The experimental therapy uses a patient's own tumor lysate and white blood cells from which precursors of the dendritic cells are isolated. The dendritic cell is the starter engine of the immune system. The white cells are then made into dendritic cells and they are educated to "teach" the immune system how to recognize brain cancer cells. Eligible patients will receive a series of injections of DCVax-L, to activate and then boost the immune response to the tumor cells.

The primary study endpoint is OS (overall survival) compared to external controls in newly diagnosed glioblastoma, and the first secondary endpoint is OS compared to external controls in recurrent glioblastoma.

Side effects reported from early trials are mostly mild, and may include skin reactions of redness, pain & swelling at the injection site.

ELIGIBILITY:
Inclusion Criteria:

All patients must meet the following inclusion criteria. All tests and eligibility criteria must be completed within four weeks of completion of radiation and chemotherapy, following surgery.

* Patients must have sufficient tumor lysate protein that was generated from the surgically obtained tumor material. Patients must also have sufficient DCVax-L product available after manufacturing. These determinations will be made by Cognate BioServices, Inc. (Cognate) and communicated to the clinical site through the Sponsor, or its designee.
* Patients with newly diagnosed, unilateral GBM (Grade IV) are eligible for this protocol. An independent neuropathologist will review this diagnosis during the enrollment process.
* Subjects ≥18 and ≤70 years of age at surgery who are capable of informed consent. Patients must be able to understand and sign the informed consent documents indicating that they are aware of the investigational nature of this study.
* Patients must have a life expectancy of >8 weeks.
* Patients must have a KPS rating of ≥70 at the baseline visit (Visit 3).
* Primary therapy must consist of surgical resection with the intent for a gross or near total resection of the contrast-enhancing tumor mass, followed by conventional external beam radiation therapy and concurrent Temodar chemotherapy. Patients having a biopsy only will be excluded. These primary treatments must be completed at least two weeks prior to first immunization.
* Patients may have received steroid therapy as part of their primary treatment. Steroid treatment must be stopped at least 10 days prior to leukapheresis.
* Patients must not have progressive disease at completion of radiation therapy. Patients with suspected pseudoprogression will be enrolled and analyzed separately.
* Patients must be willing to forego cytotoxic anti-tumor therapies except temozolomide essentially according to the schedule of the Stupp Protocol (Stupp et al. N Engl J Med 352: 987-96, 2005) while being treated with DCVax-L. DCVax-L treatment must be given as described and temozolomide/Temodar treatment schedules must be given essentially according to the Stupp Protocol.
* Patients must have adequate bone marrow function (e.g., hemoglobin >10 g/dl, white blood count 3600-11,000mm3, absolute granulocyte count ≥1,500/mm3, absolute lymphocyte count ≥1,000/mm3, and platelet count ≥100K/mm3. Eligibility level of hemoglobin can be reached by transfusion.
* Adequate liver function (SGPT, SGOT, and alkaline phosphatase ≤1.5 times upper limits of normals (ULN) and total bilirubin ≤1.5mg/dl), and adequate renal function (BUN or creatinine ≤1.5 times ULN) prior to starting therapy.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 348 (Estimated)
Dates: Start 2006-12; Primary Completion 2022-11 (Estimated)

PRIMARY OUTCOMES:
The primary objective of this study is to compare overall survival (OS) between patients randomized to DCVax-L and control patients from comparable, contemporaneous trials who received standard of care therapy only, in newly diagnosed glioblastoma. | Until death

SECONDARY OUTCOMES:
The first secondary objective is to compare overall survival (OS) between patients randomized to placebo who received DCVax-L treatment following disease recurrence, and control patients from comparable, contemporaneous clinical trials, in recurrent GBM. | Until death

CONTACTS AND LOCATIONS:
Overall Officials: Linda Liau, M.D., Principal Investigator — University of California, Los Angeles; Marnix L. Bosch, MBA, PhD, Study Director — Northwest Biotherapeutics
Locations (86):
- United States (71):
  - University of Alabama at Birmingham, Birmingham, Alabama
  - University of Arkansas for Medical Sciences, Little Rock, Arkansas
  - Sutter East Bay Neuroscience Institute-Eden Medical Center, Castro Valley, California
  - City of Hope, Duarte, California
  - UCSD Moores Cancer Center, La Jolla, California
  - Kaiser Permanente - Los Angeles, Los Angeles, California
  - UCLA Medical Center, Los Angeles, California
  - Hoag Memorial Hospital Presbyterian, Newport Beach, California
  - St. Joseph Hospital of Orange, Orange, California
  - University of California, Irvine Medical Center, Orange, California
  - Kaiser Permanente - Redwood City, Redwood City, California
  - Sutter Institute for Medical Research, Sacramento, California
  - University of Colorado Cancer Center, Aurora, Colorado
  - Colorado Neurological Institute, Englewood, Colorado
  - Georgetown University Medical Center, Washington D.C., District of Columbia
  - University of Florida, Gainesville, Florida
  - Memorial Cancer Institute, Hollywood, Florida
  - Mount Sinai Community Clinical Oncology Program, Miami Beach, Florida
  - Moffitt Cancer Center, Tampa, Florida
  - Piedmont Atlanta Hospital, Atlanta, Georgia
  - Rush University Medical Center, Chicago, Illinois
  - Illinois Cancer Care, Peoria, Illinois
  - Cadence Cancer Center, Warrenville, Illinois
  - IU Simon Cancer Center, Indianapolis, Indiana
  - University of Kansas Cancer Center, Westwood, Kansas
  - Markey Cancer Center/University of Kentucky, Lexington, Kentucky
  - Norton Cancer Institute, Louisville, Kentucky
  - Tufts Medical Center, Boston, Massachusetts
  - Beth Israel Deaconess Medical Center, Boston, Massachusetts
  - University of Michigan Cancer Center, Ann Arbor, Michigan
  - Henry Ford Hospital, Detroit, Michigan
  - Spectrum Health, Grand Rapids, Michigan
  - John Nasseff Neuroscience Institute at Abbott Northwestern Hospital, Minneapolis, Minnesota
  - St. Luke's Hospital, Kansas City, Missouri
  - Washington University School of Medicine, St Louis, Missouri
  - The Brain Tumor Center at JFK Medical Center, Edison, New Jersey
  - John Theurer Cancer Center at Hackensack University Medical Center, Hackensack, New Jersey
  - The Valley Hospital, Ridgewood, New Jersey
  - Overlook Hospital, Summit, New Jersey
  - Capital Health Regional Medical Center, Trenton, New Jersey
  - Long Island Brain Tumor Center at Neurological Surgery, P.C., Lake Success, New York
  - North Shore University Hospital, Manhasset, New York
  - New York University Clinical Cancer Center, New York, New York
  - Mount Sinai Medical Center, New York, New York
  - Columbia University Medical Center, New York, New York
  - University of Rochester Medical Center, Rochester, New York
  - Stony Brook Medicine, Stony Brook, New York
  - Brain and Spine Surgeons of New York and Northern Westchester Hospital, White Plains, New York
  - University of North Carolina, Chapel Hill, Chapel Hill, North Carolina
  - Wake Forest Baptist Medical Center, Winston-Salem, North Carolina
  - University of Cincinnati Cancer Institute, Cincinnati, Ohio
  - University Hospitals Seidman Cancer Center, Cleveland, Ohio
  - Cleveland Clinic Foundation, Cleveland, Ohio
  - Ohio State University, Columbus, Ohio
  - OhioHealth, Columbus, Ohio
  - Oklahoma University Health Science Center, Oklahoma City, Oklahoma
  - Geisinger Medical Center, Danville, Pennsylvania
  - Hospital of the University of Pennsylvania, Philadelphia, Pennsylvania
  - Jefferson Hospital for Neuroscience, Philadelphia, Pennsylvania
  - Temple University School of Medicine, Philadelphia, Pennsylvania
  - Rhode Island Hospital, Providence, Rhode Island
  - Medical University of South Carolina Hospitals and Clinics, Charleston, South Carolina
  - Saint Thomas Research Institute, Nashville, Tennessee
  - Vanderbilt Ingram Cancer Center, Nashville, Tennessee
  - Baylor Research Institute, Dallas, Texas
  - The Methodist Hospital, Houston, Texas
  - University of Texas Health Science Center at Houston, Houston, Texas
  - Cancer Therapy & Research at University of Texas Health Science Center San Antonio, San Antonio, Texas
  - Benaroya Research Institute at Virginia Mason, Seattle, Washington
  - Swedish Hospital Neuroscience Research, Seattle, Washington
  - Aurora Saint Luke's Medical Center, Milwaukee, Wisconsin
- Canada (2):
  - Montreal Neurological Institute, McGill University, Montreal, Quebec
  - CHUS - Hôpital Fleurimont, Sherbrooke, Quebec
- Germany (9):
  - Universitätsklinikum Heidelberg Neurochirurgische Klinik, Heidelberg, Baden-Wurttemberg
  - Katharinenhospital, Stuttgart, Baden-Wurttemberg
  - Universitätsklinikum FrankfurtKlinik und Poliklinik für Neurochirurgie, Frankfurt am Main, Hesse
  - Universitätsklinikum Bonn Nervenklinik (Zentrum), Klinik und Poliklinik für Neurochirurgie, Bonn, North Rhine-Westphalia
  - Universitätsklinikum Klinik für allgemeine Neurochirurgie, Cologne, North Rhine-Westphalia
  - Klinik für Neurochirurgie, Klinikum Chemnitz gGmbH, Chemnitz, Saxony
  - Universitätsklinikum Carl Gustav Carus an der Technischen Universität Dresden, Dresden, Saxony
  - BG-Kliniken Bergmannstrost, Klinik für Neurochirurgie, Halle, Saxony-Anhalt
  - Neurochirurgische Klinik, Hamburg
- United Kingdom (4):
  - Addenbrookes NHS Trust, Cambridge, Cambridgeshire, East Anglia
  - Kings College Hosital NHS Foundation Trust, London, Greater London
  - University College Hospital London, London, Greater London
  - University Hospital of Birmingham NHS Foundation Trust, Birmingham, West Midlands

REFERENCES:
- [Derived] Liau LM, Ashkan K, Brem S, Campian JL, Trusheim JE, Iwamoto FM, Tran DD, Ansstas G, Cobbs CS, Heth JA, Salacz ME, D'Andre S, Aiken RD, Moshel YA, Nam JY, Pillainayagam CP, Wagner SA, Walter KA, Chaudhary R, Goldlust SA, Lee IY, Bota DA, Elinzano H, Grewal J, Lillehei K, Mikkelsen T, Walbert T, Abram S, Brenner AJ, Ewend MG, Khagi S, Lovick DS, Portnow J, Kim L, Loudon WG, Martinez NL, Thompson RC, Avigan DE, Fink KL, Geoffroy FJ, Giglio P, Gligich O, Krex D, Lindhorst SM, Lutzky J, Meisel HJ, Nadji-Ohl M, Sanchin L, Sloan A, Taylor LP, Wu JK, Dunbar EM, Etame AB, Kesari S, Mathieu D, Piccioni DE, Baskin DS, Lacroix M, May SA, New PZ, Pluard TJ, Toms SA, Tse V, Peak S, Villano JL, Battiste JD, Mulholland PJ, Pearlman ML, Petrecca K, Schulder M, Prins RM, Boynton AL, Bosch ML. Association of Autologous Tumor Lysate-Loaded Dendritic Cell Vaccination With Extension of Survival Among Patients With Newly Diagnosed and Recurrent Glioblastoma: A Phase 3 Prospective Externally Controlled Cohort Trial. JAMA Oncol. 2023 Jan 1;9(1):112-121. doi: 10.1001/jamaoncol.2022.5370. PMID 36394838
- [Derived] Liau LM, Ashkan K, Tran DD, Campian JL, Trusheim JE, Cobbs CS, Heth JA, Salacz M, Taylor S, D'Andre SD, Iwamoto FM, Dropcho EJ, Moshel YA, Walter KA, Pillainayagam CP, Aiken R, Chaudhary R, Goldlust SA, Bota DA, Duic P, Grewal J, Elinzano H, Toms SA, Lillehei KO, Mikkelsen T, Walbert T, Abram SR, Brenner AJ, Brem S, Ewend MG, Khagi S, Portnow J, Kim LJ, Loudon WG, Thompson RC, Avigan DE, Fink KL, Geoffroy FJ, Lindhorst S, Lutzky J, Sloan AE, Schackert G, Krex D, Meisel HJ, Wu J, Davis RP, Duma C, Etame AB, Mathieu D, Kesari S, Piccioni D, Westphal M, Baskin DS, New PZ, Lacroix M, May SA, Pluard TJ, Tse V, Green RM, Villano JL, Pearlman M, Petrecca K, Schulder M, Taylor LP, Maida AE, Prins RM, Cloughesy TF, Mulholland P, Bosch ML. First results on survival from a large Phase 3 clinical trial of an autologous dendritic cell vaccine in newly diagnosed glioblastoma. J Transl Med. 2018 May 29;16(1):142. doi: 10.1186/s12967-018-1507-6. PMID 29843811
- [Derived] Badhiwala J, Decker WK, Berens ME, Bhardwaj RD. Clinical trials in cellular immunotherapy for brain/CNS tumors. Expert Rev Neurother. 2013 Apr;13(4):405-24. doi: 10.1586/ern.13.23. PMID 23545055
- See also: Northwest Biotherapeutics, Inc. — http://www.nwbio.com